CLINICAL TRIAL: NCT04527796
Title: Influence of a Residential Rehabilitation Program on Body Composition in Patients with Cystic Fibrosis (children and Adults)
Brief Title: Influence of a Residential Rehabilitation Program on Body Composition in Patients with Cystic Fibrosis
Status: Terminated | Type: Observational
Why Stopped: number included
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201939582
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis
Keywords: body composition; rehabilitation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- rehabilitation: All included patients get an pre-intervention and a post intervention analysis
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — During the rehabilitation program a multidisciplinary team, consisting of a pneumologist, dietician, psychologist, social worker and several physiotherapists, coach the cystic fibrosis patients.
  The physiotherapists help with autogenic drainage and aerosol therapy (2-3 times/day) and supervise physical activity (5, 1-hour lasting, training sessions/week: swimming 2, Fitness training 2, 1 session of choice). The dietician calculates basal and theoretical energy needs . A carbohydrate-rich snack before exercise, to improve exercise tolerance and a carbohydrate-protein-rich snack afterwards to improve recuperation is provided.

SUMMARY:
The aim is to evaluate the impact of a 3-week lasting residential rehabilitation program for patients with cystic fibrosis on their nutritional status measured as BMI and body composition and pulmonary function.

DETAILED DESCRIPTION:
Cystic fibrosis Patients following a residential rehabilitation program consisting of dietary adaptation, physical therapy for airway drainage and supervised inhalation therapy and physical activity for at least 3 weeks are asked to participate. Weight, height, body composition and pulmonary function will be measured at start and end of the program. Dietary intake during the program is calculated based on a 2 day weighed intake diary and physical activity will be measured with the "SenseWear pro 3" armband.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis
* stay at the rehabilitation center for at least 3 consecutive weeks

Exclusion Criteria:

* steroid use
* absence from the program for more than 2 consecutive days

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Cystic Fibrosis
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
body composition change | day 0 and day 21 (start and end of the rehabilitation program)
  Dual energy X-ray absorptiometry measured Fat mass index (kg/m*2)
body composition change | day 0 and day 21 (start and end of the rehabilitation program)
  Dual energy X-ray absorptiometry measured fat free mass (kg/m*2)
Body mass index change | day 0 and day 21 (start and end of the rehabilitation program)
  calculated based on weight and height (kg/m*2) converted in standard deviations
Weight change | day 0 and day 21 (start and end of the rehabilitation program)
  Scale weighed weight (kg) converted in standard deviations of normal population of normal populations
pulmonary function change | day 0 and day 21 (start and end of the rehabilitation program)
  forced expiratory volume in 1 second (% of normal)
pulmonary function change | day 0 and day 21 (start and end of the rehabilitation program)
  Forced Vital capacity (% of normal)

SECONDARY OUTCOMES:
Physical activity | Week 1
  "SenseWear pro 3" armband measured physical activity
dietary intake | 2 days/week for 3 consecutive weeks
  macronutrient intake measured based on 2 days/week weighed nutritional intake

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Van Biervliet, MD, PhD, Principal Investigator — Gent university hospital
Locations (1):
- Zeepreventorium de Haan, De Haan, Belgium

IPD SHARING:
Plan to Share IPD: No